CLINICAL TRIAL: NCT01070979
Title: A Multicenter, Double-Blind, Controlled, Randomized Study to Compare the Efficacy in Relief of Hot Flushes in Women Receiving Oral Estradiol Acetate Tablets, Oral Estradiol Tablets or Oral Conjugated Equine Estrogens
Brief Title: Hormone Replacement Therapy for Use in Postmenopausal Women for Relief of Hot Flushes and Urogenital Symptoms.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-03602.1
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Results first posted 2011-04-08 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Hormone Replacement Therapy
MeSH Terms: interventions — Estradiol; Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Estradiol acetate (E3A) (Experimental)
  Interventions: Drug: Estradiol acetate
- Estradiol (Active Comparator)
  Interventions: Drug: Estradiol
- Conjugated equine estrogens (CEE): (Active Comparator)
  Interventions: Drug: Conjugated equine estrogens

INTERVENTIONS:
Drug: Estradiol acetate — Tablet containing 0.9 mg E3A, daily oral administration.
  Arms: Estradiol acetate (E3A)
Drug: Estradiol — Tablet containing 1 mg estradiol, daily oral administration.
  Other Names: Estrace
  Arms: Estradiol
Drug: Conjugated equine estrogens — Tablet containing 0.625 mg CEE, daily oral administration.
  Other Names: Premarin
  Arms: Conjugated equine estrogens (CEE):

SUMMARY:
Multicenter, double-blind, controlled, parallel group, randomized study to compare the clinical benefit of Estradiol acetate tablets, estradiol tablets and conjugated equine estrogen tablets, each administered orally, once daily, to postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years of age; bilateral oophorectomy ≥ 35 years of age.
2. Non-hysterectomized women:

   * Amenorrhea for ≥ 12 months or
   * Amenorrhea for ≤ 12 months, but longer than 6 months, and serum FSH (follicle stimulating hormone) levels > 40 units/L and serum estradiol levels < 20 pg /mL,

   Hysterectomized women:
   * Bilateral oophorectomy - subjects may enter the study 6 weeks after surgery or
   * History of removal of ovaries may be confirmed by - serum FSH levels > 40 units/L and serum estradiol levels < 20 pg/mL or via surgical report / ultrasound.
3. Seven or more moderate or severe hot flushes daily for 1 week or 60 or more moderate or severe flushes in 1 week during the 2 week screening period prior to study entry.

Exclusion Criteria:

1. Hormone therapy administered via the following routes and during the specified timeframes: oral within 8 weeks, vaginal (rings, creams, gels) within 1 week, transdermal within 4 weeks, intramuscular within 6 weeks, progestational implants, estrogen or estrogen/progestational injectable drug therapy within 3 months, estrogen pellet or progestational injectable within 6 months.
2. Abnormal Pap smear suggestive of low grade squamous intraepithelial lesion (LGSIL) or worse. Enrollment of subjects with an ASCUS (atypical squamous cells of undetermined significance) interpretation must be discussed with the sponsor prior to randomization.
3. Urinary tract infection
4. Congestive heart failure
5. Uncontrolled hypertension; sitting systolic BP ≥ 160 mmHg or diastolic ≥ 95 mmHg
6. History of stroke or transient ischemic attacks
7. Treatment with anticoagulants (heparin or warfarin).
8. Uncontrolled thyroid disorders.
9. Insulin-dependent diabetes mellitus.
10. Increase frequency or severity of headaches including migraines during previous estrogen therapy.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2003-02; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Warner Chilcott
Locations (31):
- United States (31):
  - Warner Chilcott Investigational Site, Phoenix, Arizona
  - Warner Chilcott Investigational Site, Carmichael, California
  - Warner Chilcott Investigational Site, San Diego, California
  - Warner Chilcott Investigational Site, Aventura, Florida
  - Warner Chilcott Investigational Site, Boynton Beach, Florida
  - Warner Chilcott Investigational Site, Clearwater, Florida
  - Warner Chilcott Investigational Site, Daytona Beach, Florida
  - Warner Chilcott Investigational Site, Gainesville, Florida
  - Warner Chilcott Investigational Site, Longwood, Florida
  - Warner Chilcott Investigational Site, Melbourne, Florida
  - Warner Chilcott Investigational Site, Miami, Florida
  - Warner Chilcott Investigational Site, Palm Springs, Florida
  - Warner Chilcott Investigational Site, Pinellas Park, Florida
  - Warner Chilcott Investigational Site, Sarasota, Florida
  - Warner Chilcott Investigational Site, Venice, Florida
  - Warner Chilcott Investigational Site, Roswell, Georgia
  - Warner Chilcott Investigational Site, Chicago, Illinois
  - Warner Chilcott Investigational Site, Peoria, Illinois
  - Warner Chilcott Investigational Site, Laurel, Maryland
  - Warner Chilcott Investigational Site, Lincoln, Nebraska
  - Warner Chilcott Investigational Site, Raleigh, North Carolina
  - Warner Chilcott Investigational Site, Winston-Salem, North Carolina
  - Warner Chilcott Investigational Site, Cleveland, Ohio
  - Warner Chilcott Investigational Site, Columbus, Ohio
  - Warner Chilcott Investigational Site, Mogadore, Ohio
  - Warner Chilcott Investigational Site, Portland, Oregon
  - Warner Chilcott Investigational Site, Pittsburgh, Pennsylvania
  - Warner Chilcott Investigational Site, Nashville, Tennessee
  - Warner Chilcott Investigational Site, Salt Lake City, Utah
  - Warner Chilcott Investigational Site, Spokane, Washington
  - Warner Chilcott Investigational Site, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of postmenopausal women for relief of hot flushes and urogenital symptoms beginning Feb '03 at 33 sites in the US.
Pre-assignment Details: Discontinue estrogen/hormone therapy prior to enrollment
Groups:
- Estradiol Acetate (E3A): 1 tablet daily containing 0.9 mg estradiol acetate
- Estradiol: 1 tablet daily containing 1 mg estradiol
- Conjugated Equine Estrogens (CEE): 1 tablet daily containing 0.625 mg conjugated equine estrogen
Period: Overall Study
Arm/Group | Estradiol Acetate (E3A) | Estradiol | Conjugated Equine Estrogens (CEE)
Started | 79 | 85 | 85
Completed | 68 | 73 | 72
Not Completed | 11 | 12 | 13
Not completed — Adverse Event | 2 | 3 | 3
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Protocol Violation | 0 | 2 | 6
Not completed — Surgery, moving, personal, abn. labs | 4 | 4 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — No study drug taken | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol Acetate (E3A) | Estradiol | Conjugated Equine Estrogens (CEE) | Total
Number analyzed (Participants) | 79 | 85 | 85 | 249
Age Continuous [Mean (Standard Deviation); unit: years] | 52.2 (6.6) | 52.3 (7.0) | 53.8 (6.3) | 52.8 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 85 | 85 | 249
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 79 | 85 | 85 | 249

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Number of Moderate to Severe Hot Flushes, Week 4, ITT (Intention to Treat) Population
Description: Severity of hot flush definitions: mild - sensation of heat without perspiration, moderate - sensation of heat with perspiration, able to continue activity, severe - sensation of heat with perspiration, causing the subject to stop activity or awaken from sleep
Time Frame: Baseline to Week 4
Population: Intention to Treat (ITT) with Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Change in Hot Flush Count
Arm/Group | Estradiol Acetate (E3A) | Estradiol | Conjugated Equine Estrogens (CEE)
Number analyzed (Participants) | 77 | 80 | 84
Change in Hot Flush Count | -54.1 (4.5) | -62.0 (4.5) [0.721 to 1.048] | -54.5 (4.3) [0.833 to 1.178]

2. Secondary Outcome: Mean Change From Baseline in the Severity of Moderate to Severe Hot Flushes, Week 4, ITT Population
Description: Patient self-reported outcome. Severity of hot flush definitions: mild (1) - sensation of heat without perspiration, moderate (2) - sensation of heat with perspiration, able to continue activity, severe (3) - sensation of heat with perspiration, causing the subject to stop activity or awaken from sleep. Minimum 0/no hot flushes, Maximum 3/all severe hot flushes. Lower the score the greater the improvement in reducing hot flushes.
Time Frame: Baseline to Week 4
Population: Intention to Treat (ITT) with Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Change in Score
Arm/Group | Estradiol Acetate (E3A) | Estradiol | Conjugated Equine Estrogens (CEE)
Number analyzed (Participants) | 77 | 80 | 84
Change in Score | -0.53 (0.106) | -0.51 (0.106) | -0.59 (0.102)

3. Primary Outcome: Mean Change From Baseline in the Number of Moderate to Severe Hot Flushes, Week 12, ITT Population
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: Intention to Treat (ITT) with Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Change in Hot Flush Count
Arm/Group | Estradiol Acetate (E3A) | Estradiol | Conjugated Equine Estrogens (CEE)
Number analyzed (Participants) | 77 | 80 | 84
Change in Hot Flush Count | -63.6 (4.8) | -72.2 (4.7) | -67.2 (4.6)

4. Secondary Outcome: Mean Change From Baseline in the Severity of Moderate to Severe Hot Flushes, Week 12, ITT Population
Description: as for outcome 2
Time Frame: Baseline to Week 12
Population: Intention to Treat (ITT) with Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Change in Score
Arm/Group | Estradiol Acetate (E3A) | Estradiol | Conjugated Equine Estrogens (CEE)
Number analyzed (Participants) | 77 | 80 | 84
Change in Score | -1.05 (0.127) | -1.34 (0.125) | -1.17 (0.122)

5. Secondary Outcome: Mean Change From Baseline in Total Urogenital Symptom Score, Week 4, ITT Population
Description: Urogenital Symptom Severity scored none=0, mild=1, moderate=2, severe=3.
Time Frame: Baseline to Week 4
Population: Intention to Treat (ITT) with Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Change in Score
Arm/Group | Estradiol Acetate (E3A) | Estradiol | Conjugated Equine Estrogens (CEE)
Number analyzed (Participants) | 77 | 80 | 84
Change in Score | -1.89 (0.413) | -2.26 (0.407) | -1.96 (0.398)

6. Secondary Outcome: Change From Baseline in Total Urogenital Symptom Score, Week 8, ITT Population
Description: Urogenital Symptom Severity scored none=0, mild=1, moderate=2, severe=3.
Time Frame: Baseline to Week 8
Population: Intention to Treat (ITT) with Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Change in Score
Arm/Group | Estradiol Acetate (E3A) | Estradiol | Conjugated Equine Estrogens (CEE)
Number analyzed (Participants) | 77 | 80 | 84
Change in Score | -1.96 (0.432) | -2.58 (0.425) | -2.42 (0.416)

7. Secondary Outcome: Change From Baseline in Total Urogenital Symptom Score, Week 12, ITT Population
Description: Urogenital Symptom Severity scored none=0, mild=1, moderate=2, severe=3.
Time Frame: Baseline to Week 12
Population: Intention to Treat (ITT) with Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Change in Score
Arm/Group | Estradiol Acetate (E3A) | Estradiol | Conjugated Equine Estrogens (CEE)
Number analyzed (Participants) | 77 | 80 | 84
Change in Score | -2.49 (0.437) | -2.59 (0.431) | -2.52 (0.422)

ADVERSE EVENTS:
Time Frame: 7 months
Description: February 2003 thru September 2003, One subject randomized to estradiol group never took any study drug therefore not included in AE assessment.
Arm/Group | Estradiol Acetate (E3A) | Estradiol | Conjugated Equine Estrogens (CEE)
Serious Adverse Events (participants affected / at risk) | 0/79 | 1/84 | 0/85
Other Adverse Events (participants affected / at risk) | 19/79 | 25/84 | 30/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol Acetate (E3A) (N=79) | Estradiol (N=84) | Conjugated Equine Estrogens (CEE) (N=85)
metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Estradiol Acetate (E3A) (N=79) | Estradiol (N=84) | Conjugated Equine Estrogens (CEE) (N=85)
Breast Tenderness (Reproductive system and breast disorders) | 2 | 5 | 5
Nausea (Gastrointestinal disorders) | 4 | 1 | 2
Headache (Nervous system disorders) | 3 | 5 | 6
Metrorrhagia (Reproductive system and breast disorders) | 2 | 3 | 4
Abdominal Distention (Gastrointestinal disorders) | 1 | 4 | 2
Vaginosis Fungal (Infections and infestations) | 0 | 1 | 3
Weight Increased (Investigations) | 1 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Nasopharyngitis (Nervous system disorders) | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less